CLINICAL TRIAL: NCT01661244
Title: A Randomised, Double-blind, Placebo-controlled, Two Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Treatment With Single and Repeat Doses of Inhaled RV568 in Healthy Volunteers
Brief Title: A Study to Investigate the Safety and Tolerability of a New Inhaled Formulation of RV568 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVH007
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: COPD; Healthy Volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A - Single dose escalation (Experimental)
  Interventions: Drug: RV568 single dose; Drug: RV568 matching placebo single dose
- Part B - 14 day repeat dose escalation (Experimental)
  Interventions: Drug: RV568 repeat dose; Drug: RV568 matching placebo repeat dose

INTERVENTIONS:
Drug: RV568 single dose — Safety and tolerability of single escalating doses in normal human volunteers
  Arms: Part A - Single dose escalation
Drug: RV568 matching placebo single dose — Safety and tolerability of escalating repeat doses in normal human volunteers.
  Arms: Part A - Single dose escalation
Drug: RV568 repeat dose — Safety and tolerability of escalating repeat doses in normal human volunteers.
  Arms: Part B - 14 day repeat dose escalation
Drug: RV568 matching placebo repeat dose — Safety and tolerability of escalating repeat doses in normal human volunteers.
  Arms: Part B - 14 day repeat dose escalation

SUMMARY:
RV568 is being developed as a possible treatment of smoking related lung disease (also known as Chronic Obstructive Pulmonary Disease - COPD).

The main purpose of this study is to examine the safety and tolerability of a new inhaled formulation of RV568 in healthy volunteers. The study will be run in two parts; Part A and Part B. Part A (Cohorts 1, 2 & 3) will investigate 6 different dose levels of RV568 given as a single dose and Part B (Cohorts 4 & 5) will investigate 2 different dose levels of RV568 given once a day for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a physician, based on a full medical evaluation including medical history, physical examination, and laboratory tests.
* Body weight ≥50 kg and body mass index within the range 19-29 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTc(B) or QTc(F) <450 msec (or QTc <480 msec in healthy subjects with right bundle branch block).
* Capable of complying with all study restrictions and procedures including ability to use the Dry Powder Inhaler correctly.
* Spirometry readings (FEV1 and FVC) to be ≥ 80% predicted value and FEV1/FVC ratio > 0.7 calculated using ECCS reference equations.
* Vital sign assessments within normal ranges (systolic blood pressure (SBP) 90 140 mm/Hg; diastolic blood pressure (DBP) 55 - 90 mm/Hg; heart rate (HR) 40 - 100 bpm).
* Agree not to use prescription medications within 14 days before first administration of study medication and through the duration of the study (with the exception of contraception and hormone replacement therapy (HRT)).
* Agree not to use over the counter (OTC) medications (including corticosteroids, decongestants, antihistamines, aspirin and other non-steroidal anti-inflammatory drugs (NSAIDs)) and herbal medication (including, but not limited to, herbal tea and St. John's Wort), within 14 days before first administration of study medication and through to the final follow up visit, unless approved by the Investigator and Sponsor Medical Monitor. Occasional use of paracetamol at recommended doses (≤ 1 g/ 6 hours and ≤ 2 g/day) and continued pre-existing use of vitamins at recommended doses is allowed.

Exclusion Criteria:

* Any acute or chronic illness or clinically relevant abnormality identified on the screening medical assessment, laboratory tests or ECG.
* Upper or lower respiratory tract infection within 4 weeks of the screening visit.
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Positive urinary drugs or breath alcohol test at screening or prior to dosing.
* The Investigator suspects drug or alcohol abuse.
* A positive test for human immunodeficiency virus antibody.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in any other study of an investigational drug during the 3 months before receipt of the first dose of study medication or has previously received RV568.
* Regular use of prescription or non-prescription drugs within 14 days prior to the first dose of study medication.
* Allergy to any of the active or inactive ingredients in the study medication.
* History of drug, or other allergy that, in the opinion of the Investigator or Sponsor Medical Monitor, would contraindicate their participation.
* The subject is a smoker (regular or irregular), or has smoked or used nicotine-containing products within the 6 months prior to screening.
* Positive carbon monoxide breath test at the screening visit indicative of smoking or use of tobacco or nicotine-containing products.
* Donation of blood in excess of 500 mL within a 3 month period prior to screening, or if study participation would result in blood loss in excess of 500 mL in a 3 month period.
* The subject is unable or unwilling to comply fully with the study protocol.
* Subject is mentally or legally incapacitated.
* Subject is an employee of the Sponsor or contract research organization (CRO), or a relative of an employee of the Sponsor or CRO.
* Unable or unwilling to undergo multiple venepuncture procedures or the subject has poor access to veins suitable for cannulation.
* A positive pregnancy test or is a lactating (nursing) female.
* Any other reason that the Investigator considers makes the subject unsuitable to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Cohort 1, 56 days; Cohorts 2 & 3, 28 days; Cohorts 4 & 5, 35 days
  Assessment of the number of adverse events reported by subjects following dosing.
ECG assessment | Cohort 1, 56 days; Cohorts 2 & 3, 28 days; Cohorts 4 & 5, 35 days
  Change from pre-dose values.
Vital signs assessment | Cohort 1, 56 days; Cohorts 2 & 3, 28 days; Cohorts 4 & 5, 35 days
  Change from pre-dose values
Spirometry assessment | Cohort 1, 56 days; Cohorts 2 & 3, 28 days; Cohorts 4 & 5, 35 days
  Change from pre-dose values

SECONDARY OUTCOMES:
Plasma RV568 levels | Cohorts 1, 2 & 3: Day 1 (0, 15, 30 & 45 min and 1, 2, 4, 6, 8, 10, 12 and 24 h), then 7, 14 and 28 days. Cohorts 4 & 5: Day 1, 7 & 14 (0, 15, 30 & 45 min and 1, 2, 4, 6, 8, 10, 12 and 24 h), Day 10, 11, 12 & 13 (0 & 30 min), then Day 21, 28 and 35

CONTACTS AND LOCATIONS:
Overall Officials: Dr Garth Rapeport, Study Director — Respivert Ltd
Locations (1):
- London, United Kingdom